CLINICAL TRIAL: NCT02832804
Title: Effect of Transcranial Direct-current Stimulation Therapy on Primary Chronic Insomnia Patients: A Pilot Study.Insomnia Patients
Brief Title: Effect of Transcranial Direct-current Stimulation Therapy on Primary Chronic Insomnia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ki-Young Jung, professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1509-061-703
Record Dates: First submitted 2016-04-18; First posted 2016-07-14 (Estimated); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Primary Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- anodal stimulation (Experimental): 10 person The patients treated by anodal stimulation (2mA) for 20 minutes
  Interventions: Device: transcranial Direct Current Stimulation
- cathodal stimulation (Active Comparator): 10 person The patients treated by cathodal stimulation (1-2mA) for 20 minutes
  Interventions: Device: transcranial Direct Current Stimulation
- sham stimulation (Sham Comparator): 10 person The patients treated by anodal stimulation (1-2mA) for 15 seconds
  Interventions: Device: transcranial Direct Current Stimulation

INTERVENTIONS:
Device: transcranial Direct Current Stimulation — Experimental: anodal stimulation (2mA) for 20 minutes Active Comparator: cathodal stimulation (2mA) for 20 minutes Sham Comparator: sham stimulation (2mA) for 15 seconds
  Other Names: HDCstim (direct current stimulator)

SUMMARY:
To evaluate the clinical efficacy and safety of neuromodulation by transcranial direct current stimulation (tDCS) in the patients with primary chronic insomnia .

DETAILED DESCRIPTION:
* visit 1

  * to fill in a questionnaire (Clinical Global Impression, CGI; Leeds Sleep Evaluation Questionnaire, LSEQ; Stanford Sleepiness Scale, SSS; Hospital Anxiety and Depression Scale, HADS; 36-Item Short Form Survey, SF-36)
  * EEG
* visit 2-6

  * tDCS stimulation (monday ~ friday)
  * anodal / cathodal / sham
  * to fill in a questionnaire (CGI, LSEQ, SSS, HADS)
  * analysis the results of sleep log and actigraphy
* visit 7 : 1 week after treatment

  * to fill in a questionnaire (CGI, LSEQ, SSS, HADS)
  * analysis the results of sleep log and actigraphy
  * EEG
* visit 8 : 1 month after treatment

  * to fill in a questionnaire (CGI, LSEQ, SSS, HADS, SF-36)
  * analysis the results of sleep log

ELIGIBILITY:
Inclusion Criteria:

* adult (older than 19 years)
* primary insomnia
* right handed
* agree with participation of this study

Exclusion Criteria:

* diagnosed with epilepsy or history of seizure
* change of antipsychotic drug within 1 month
* under suspicion of sleep apnea or periodic limb movement disorder
* mental retardation (IQ < 70)
* pregnant woman

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
sleep log and actiwatch | Change from baseline at 1 week
  Changes of sleep quality

SECONDARY OUTCOMES:
questionnaire | Change from baseline at 1 month
EEG spectrum analysis | Change from baseline at 1 month
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Change from baseline at 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Ki-Young Jung, professor, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided